CLINICAL TRIAL: NCT02550964
Title: Incidence and Risk Factor Evaluation for Toxic Maculopathy Associated With Hydroxychloroquine and Chloroquine
Brief Title: Incidence and Risk Factor of Hydroxychloroquine and Chloroquine Retinopathy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, JooYong Lee, Associate Professor, Asan Medical Center
Other Study IDs: 2013-0826
Record Dates: First submitted 2015-09-14; First posted 2015-09-16 (Estimated); Last update posted 2015-09-18 (Estimated); Status verified 2015-09

CONDITIONS: Toxic Maculopathy
Keywords: Autoimmune Disease; Rheumatoid Arthritis; Systemic Lupus Erythematosus; Hydroxychloroquine(HCQ); Chloroquine(CQ); Toxic Maculopathy
MeSH Terms: conditions — Autoimmune Diseases; Arthritis, Rheumatoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HCQ/CQ: Patients who treated with HCQ(Hydroxychloroquine) or CQ(Chloroquine) for autoimmune diseases such as Rheumatoid arthritis(RA), systemic lupus erythematosus(SLE) will be recruited, and get the composite examination for toxic maculopathy.
  Interventions: Procedure: Composite Examination

INTERVENTIONS:
Procedure: Composite Examination — First, patients will get the baseline ophthalmologic exam and medical evaluation by physicians. As a diagnostic method, the composite examination including fundus photography, fundus autofluorescence, spectral-domain optical coherence tomography, Humphrey visual field test and multifocal electroretinography will be tested once every year.

SUMMARY:
The purpose of this study is to evaluate the incidence and risk factor of toxic maculopathy who treated with hydroxychloroquine or chloroquine due to their autoimmune disease such as rheumatoid arthritis or systemic lupus erythematosus. Total 5-year of the study periods, the investigators will screen these patients by baseline examination (Fundus photography, fundus autofluorescence, spectral-domain optical coherence tomography, Humphrey visual field test and multifocal electroretinography) and observe with same examination for every year.

ELIGIBILITY:
Inclusion Criteria:

* Patient who treated with HCQ or CQ due to autoimmune diseases such as RA, SLE
* Patient who did not previously diagnosed with HCQ/CQ toxic retinopathy

Exclusion Criteria:

* Aged less than 19 years

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The purpose of this cohort study is to evaluate the incidence and risk factor. We will recruit a total of 124 participants considering the study budget.
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxic maculopathy associated with HCQ or CQ | 1 years

SECONDARY OUTCOMES:
Risk factor of HCQ/CQ retinopathy | 5 years
Characteristics and type of HCQ/CQ retinopathy (parafoveal or pericentral retinopathy) | 5 years
Progression of retinopathy after drug cessation | 1 years

CONTACTS AND LOCATIONS:
Overall Officials: JooYong Lee, Professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea